CLINICAL TRIAL: NCT00008138
Title: Phase II Evaluation Of Neoadjuvant Chemotherapy, Interval Debulking Followed By Intraperitoneal Chemotherapy In Women With Stage III And IV Epithelial Ovarian Cancer, Fallopian Tube Cancer Or Primary Peritoneal Cancer
Brief Title: S0009 Combination Chemo and Surgery in Stage III or Stage IV Ovarian Cancer
Acronym: S0009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068380; U10CA032102 (NIH); S0009 (Other: SWOG)
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Paclitaxel; Cytoreduction Surgical Procedures; Surgical Procedures, Operative; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemo/debulking surgery/IP chemo (Experimental): neoadjuvant chemotherapy (carboplatin and paclitaxel) followed by debulking surgery followed by intraperitoneal chemotherapy (carboplatin and paclitaxel)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: debulking surgery

INTERVENTIONS:
Drug: carboplatin — pre-surgery - target AUC=6, Day 1 IV, q 21 days X 3 cycles post-surgery - target AUC=5, Day 1 IP, q 28 days X 6 cycles
  Other Names: carbo
Drug: paclitaxel — pre-surgery - 175 mg/m2 IV Day 1, q 21 days X 3 cycles post-surgery - 175 mg/m2 IV Day 1, q 28 days X 6 cycles AND 60 mg/m2 IP Day 8, q 28 days X 6 cycles
  Other Names: Taxol
Procedure: debulking surgery — exploratory laparotomy, interval cytoreduction (to < 1 cm residual)
  Other Names: surgery; debulking; cytoreduction; laparotomy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug or combining chemotherapy with surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and surgery in treating patients who have stage III or stage IV ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the overall survival and progression-free survival in patients with stage III or IV ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer treated with neoadjuvant paclitaxel and carboplatin followed by surgery and adjuvant paclitaxel and carboplatin.
* Estimate the percentage of these patients whose disease is successfully cytoreduced to less than 1 cm in diameter following neoadjuvant chemotherapy.
* Evaluate the toxicity of this regimen in these patients.
* Explore the relationship between tumor p53 expression, proliferation rate as measured by proliferating cell nuclear antigen and apoptotic rate, and human tumor cloning assay results at time of debulking surgery with progression-free survival and overall survival in these patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive neoadjuvant therapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Within 35 days of receiving the third course of chemotherapy, patients with at least a 50% reduction in CA 125 undergo debulking surgery. Within 35 days of undergoing surgery, patients with a tumor reduction to below 1 cm receive adjuvant therapy comprising paclitaxel IV over 3 hours followed by carboplatin intraperitoneally (IP) on day 1 and paclitaxel IP on day 8. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually for up to 5 years.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage III or IV ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer

  * Adenocarcinoma
  * Large pelvic mass and/or bulky abdominal disease and/or malignant pleural effusion
  * Pleural effusion only for stage IV (parenchymal, liver, lung, or other distant metastases not allowed)
  * No borderline or low-malignant potential tumors
* Optimal cytoreduction clinically deemed unlikely
* CA 125 at least 70 units/mL

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT no greater than 2 times ULN

Renal:

* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No congestive heart failure or cardiac arrhythmia
* No myocardial infarction or angina within past 6 months

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe gastrointestinal symptoms (i.e., partial obstruction) and/or gastrointestinal bleeding
* No grade 2 or greater sensory neuropathy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other adequately treated stage I or II cancer in complete remission
* No active or uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for this cancer

Chemotherapy:

* No prior chemotherapy for this cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior pelvic radiation for this cancer

Surgery:

* See Disease Characteristics
* Prior exploratory laparotomy allowed provided an aggressive tumor debulking procedure was not performed (e.g., bilateral salpingo-oophorectomy/total abdominal hysterectomy with omentectomy)
* Prior salpingo-oophorectomy and/or partial omentectomy allowed

Other:

* No other concurrent anti-cancer therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2001-03; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Tiersten, MD, Study Chair — NYU Langone Health

REFERENCES:
- [Result] Tiersten AD, Liu PY, Smith HO, Wilczynski SP, Robinson WR 3rd, Markman M, Alberts DS. Phase II evaluation of neoadjuvant chemotherapy and debulking followed by intraperitoneal chemotherapy in women with stage III and IV epithelial ovarian, fallopian tube or primary peritoneal cancer: Southwest Oncology Group Study S0009. Gynecol Oncol. 2009 Mar;112(3):444-9. doi: 10.1016/j.ygyno.2008.10.028. Epub 2009 Jan 12. PMID 19138791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 62 enrolled participants, 4 were deemed ineligible.
Groups:
- Experimental: Chemo/Debulking Surgery/IP Chemo: neoadjuvant chemotherapy (carboplatin and paclitaxel) followed by debulking surgery followed by intraperitoneal chemotherapy (carboplatin and paclitaxel)
Period: Neoadjuvant Chemotherapy
Arm/Group | Experimental: Chemo/Debulking Surgery/IP Chemo
Started | 58
Eligible | 58
Completed | 38
Not Completed | 20
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 6
Not completed — not protocol specified | 8
Period: Interval Debulking
Arm/Group | Experimental: Chemo/Debulking Surgery/IP Chemo
Started | 38
Received Protocol Surgery | 36
Completed | 36
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Post-Cytoreduction Chemotherapy
Arm/Group | Experimental: Chemo/Debulking Surgery/IP Chemo
Started | 26 (Among 36 patients from previous period, 5 patients rejected and 5 patients are ineligible.)
Completed | 18
Not Completed | 8
Not completed — Adverse Event | 6
Not completed — Progression | 1
Not completed — not protocol specified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Chemo/Debulking Surgery/IP Chemo
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 62 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 2
Stage [Number; unit: participants]
  Stage III | 43
  Stage IV | 15
Primary Site [Number; unit: participants]
  Ovary | 43
  Peritoneal | 14
  Not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of registration until the date of death due to any cause. Patients last known to be alive were censored at the date of last contact. Patients were followed every 3 months for the first year, every 6 months for years 2 and 3, and then annually for years 4 and 5.
Time Frame: assessed every 3 months for 1st year, then every 6 months for 2 years, then annually for years 4 and 5
Population: Only eligible patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Chemo/Debulking Surgery/IP Chemo
Number analyzed (Participants) | 58
months | 32 [22 to 37]

2. Primary Outcome: Progression-Free Survival
Description: Progression was defined as a CA-125 value that is both twice the nadir since registration and greater than 70 units/ml, and is confirmed by a second determination at least 7 days apart, or appearance of any new lesion/site. Symptomatic deterioration was defined as a global deterioration of health status requiring removal from protocol treatment. Progression-Free Survival was defined as the time from the date of registration to the date of progression, symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free were censored at last contact date.
Time Frame: Monthly during protocol treatment, then every 3 months up to the end of Year 1, then every 6 months for the next two years, then annually up to Year 5.
Population: Only eligible patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Chemo/Debulking Surgery/IP Chemo
Number analyzed (Participants) | 58
months | 21 [15 to 32]

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events every 3 weeks during neoadjuvant chemotherapy, and then every 4 weeks during intravenous/intraperitoneal chemotherapy following cytoreductive surgery.
Description: This study utilized the CTCAE (NCI Common Toxicity Criteria for Adverse Events) version 2.0
Groups:
- Neoadjuvant Paclitaxel (IV) + Carboplatin (V): Pre-surgery IV chemotherapy with paclitaxel and carboplatin
- Post-Cytoreduction Paclitaxel (IV/IP) + Carboplatin (IP): post-surgery chemotherapy with IV and IP carboplatin and paclitaxel
Arm/Group | Neoadjuvant Paclitaxel (IV) + Carboplatin (V) | Post-Cytoreduction Paclitaxel (IV/IP) + Carboplatin (IP)
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/26
Other Adverse Events (participants affected / at risk) | 41/58 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Paclitaxel (IV) + Carboplatin (V) (N=58) | Post-Cytoreduction Paclitaxel (IV/IP) + Carboplatin (IP) (N=26)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Paclitaxel (IV) + Carboplatin (V) (N=58) | Post-Cytoreduction Paclitaxel (IV/IP) + Carboplatin (IP) (N=26)
Anemia (Blood and lymphatic system disorders) | 14 (14) | 14 (14)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
PRBC transfusion (Blood and lymphatic system disorders) | 16 (16) | 3 (3)
Platelet transfusion (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Abdominal pain/cramping (Gastrointestinal disorders) | 10 (10) | 14 (14)
Constipation/bowel obstruction (Gastrointestinal disorders) | 3 (3) | 9 (9)
Diarrhea without colostomy (Gastrointestinal disorders) | 0 (0) | 7 (7)
Ileus (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 12 (12)
Vomiting (Gastrointestinal disorders) | 4 (4) | 9 (9)
Edema (General disorders) | 5 (5) | 3 (3)
Fatigue/malaise/lethargy (General disorders) | 17 (17) | 15 (15)
Fever without neutropenia (General disorders) | 5 (5) | 3 (3)
Pain-other (General disorders) | 0 (0) | 2 (2)
Allergic reaction (Immune system disorders) | 4 (4) | 0 (0)
Infection w/o 3-4 neutropenia (Infections and infestations) | 4 (4) | 0 (0)
Respiratory infect w/o neutrop (Infections and infestations) | 0 (0) | 3 (3)
Urinary tr infect w/ neutrop (Infections and infestations) | 0 (0) | 2 (2)
Urinary tr infect w/o neutrop (Infections and infestations) | 5 (5) | 0 (0)
Catheter related infection (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Local injection site reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Surgery-hemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Leukopenia (Investigations) | 9 (9) | 17 (17)
Neutropenia/granulocytopenia (Investigations) | 13 (13) | 15 (15)
SGOT (AST) increase (Investigations) | 0 (0) | 2 (2)
Thrombocytopenia (Investigations) | 7 (7) | 11 (11)
Weight loss (Investigations) | 5 (5) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 11 (11) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Dizziness/light headedness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Sensory neuropathy (Nervous system disorders) | 0 (0) | 11 (11)
Weakness (motor neuropathy) (Nervous system disorders) | 3 (3) | 2 (2)
Anxiety/agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis/embolism (Vascular disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No